CLINICAL TRIAL: NCT06519084
Title: Effect of Physical Training in Functional Capacity, Metabolic Profile, Body Composition and Quality of Life in Patients With Congenital Heart Disease
Brief Title: Home Based Program Physical Training in Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Home_based_CHD
Record Dates: First submitted 2024-02-26; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: Congenital Heart Disease; Functional Capacity; Body Composition; Quality of Life
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG - Training group (Experimental): In this group, patients were instructed to perform home-based physical training. Training was carried out 4 times a week, each exercise session lasting 40 minutes. The session consisted of aerobic exercises and muscular resistance exercises, using body weight and elastic bands.
  Interventions: Other: Home based exercise training
- CG - Control group (No Intervention): In this group, patients were advised to maintain their usual activities and not engage in physical training programs.

INTERVENTIONS:
Other: Home based exercise training — Intervention: home based physical exercise performed 4 times a week, each session lasting 40 minutes each. Aerobic and muscular resistance exercises, using body weight and elastic bands.
  The sessions were proposed through video classes, in total 12 video classes during the 12 weeks of physical training. Patients monitored their heart rate during exercise and wrote it down on spreadsheets that were monitored weekly.
  Arms: TG - Training group

SUMMARY:
Previous Studies Indicate That a Substantial Proportion of the Congenital Heart Disease Patients Has Unhealthy Lifestyle Behaviors, Such as Smoking, Lack of Physical Activity, and Inadequate Dietary Patterns, Leading to the Development of Metabolic Disorders Such as Overweight/Obesity, Metabolic Syndrome, and Chronic Diseases Such as Cardiovascular Disease. Another Highly Prevalent Risk Factor in These Patients is Sedentary Behavior; These Patients Are Not Encouraged to Engage in Sports and Exercise During Childhood Due to Their Cardiac Condition, Leading to a Progressive Decrease in Physical Capacity. Studies Have Shown That Congenital Heart Disease Patients Are Not Active Enough and That a Substantial Amount of Patients is Overweight.This Study is a Randomized Controlled Trial That Investigates the Effects of the Home Based Program Physical Training, in the Exercise Capacity, Quality of Life and Body Composition.

DETAILED DESCRIPTION:
The objective of the study was to verify the effect of home physical training on improving physical capacity, body composition, quality of life, metabolic markers in patients with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Repaired congenital heart disease of all complexities
* Age ≥ 18 years
* New York Heart Association (NYHA) Class I or II
* Able and willing to participate in a 12-week cardiac rehabilitation program

Exclusion Criteria:

* Inability to give informed consent
* Inability to participate in an exercise training program
* Severe musculoskeletal disorders.
* Patient heart failure
* Patients who perform regular physical activities.
* Patients with Univentricular Physiology,
* Patients severe asthma,
* Patients with a pacemaker.
* Patients with atrial fibrillation;
* Exercise-induced arrhythmia and/or ischemia
* Cyanosis at rest
* Severe intellectual disability

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement exercise tolerance and functional capacity (peak VO2) | Baseline to 3 months
  Change in functional capacity will be performed by cardiopulmonary exercise test and will be expressed by Peak VO2 and Predicted Peak VO2 (%). After the training program, an increase in the peak VO2(mL/kg/min) value between 10 to 15% is expected in relation to the baseline value.

SECONDARY OUTCOMES:
Change in quality of life measurement | Baseline to 3 months
  Changes in quality of life will be measure by Short Form 36 questionnaire by 8 domains: Physical functioning, Physical role functioning, body pain, general health, vitality, social functioning, emotional role functioning, mental health.
  The quality of life rating for each domain is typically measured on a scale of 0 to 100, where a score close to 100 indicates a higher or higher quality of life, while a score close to 0 suggests a lower or poorer quality of life.
Change in body composition measurement | Baseline to 3 months
  The body composition were assessment by the bioimpedance analyses in the baseline and After the home based training program with duration 12 weeks ou usual routine.
Improvement in peripheral blood flow post exercise training program | Baseline to 3 months
  Increase forearm blood flow in mL/min/100mL

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Intitute, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No